CLINICAL TRIAL: NCT06084897
Title: Radiotherapy in Patients With Metastatic Esophageal Cancer Responding to PD-1 Inhibitor Plus Chemotherapy: a Patient Preference Multicenter Randomized Phase II Trial
Brief Title: Radiotherapy in Patients With Metastatic Esophageal Cancer Responding to PD-1 Inhibitor Plus Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Anyang Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEIR 1
Record Dates: First submitted 2023-09-19; First posted 2023-10-16 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Neoplasm Metastatic; Esophageal Cancer Stage IVb
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin; Drug Therapy; Immune Checkpoint Inhibitors; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consolidation radiotherapy (Experimental): This treatment group will be receive radiotherapy on the basis of standard first-line treatment, after all planned cycles of chemotherapy combined with PD-1 inhibitor completed.
  Interventions: Drug: TP (Paclitaxel with cisplatin or carboplatin) or PF (Fluoropyrimidine with cisplatin or carboplatin) regimen depended on investigator's choice.; Biological: PD-1 inhibitor; Radiation: Consolidation Radiation
- Salvage radiotherapy (Experimental): This treatment group will be receive salvage radiotherapy on the basis of standard first-line treatment, when disease progressed and salvage radiotherapy is recommended by multidisciplinary team.
  Interventions: Drug: TP (Paclitaxel with cisplatin or carboplatin) or PF (Fluoropyrimidine with cisplatin or carboplatin) regimen depended on investigator's choice.; Biological: PD-1 inhibitor; Radiation: Salvage Radiation

INTERVENTIONS:
Drug: TP (Paclitaxel with cisplatin or carboplatin) or PF (Fluoropyrimidine with cisplatin or carboplatin) regimen depended on investigator's choice. — A maximum of six cycles was recommended for chemotherapy.
  * Fluoropyrimidine (fluorouracil or capecitabine) with carboplatin or cisplatin;
  * Paclitaxel (or Albumin-bound paclitaxel) with carboplatin or cisplatin.
  Other Names: Chemotherapy
Biological: PD-1 inhibitor — Nivolumab or Pembrolizumab or Tislelizumab or Serplulimab or Toripalimab or Sintilimab or Camrelizumab
  Other Names: Immunotherapy
Radiation: Consolidation Radiation — IMRT/VMAT technique. Patients receive radiotherapy once daily, 5 days a week for an average of 5 weeks. Radiotherapy is delivered to achieve a dosage of 49.22Gy/23f or 50Gy/25f to PGTV for lymphnode metastasis only patients and 40.66Gy/19f or 40Gy/20f for organ metastasis patients. Radiation treatment is planned after chemotherapy completed.
  Other Names: Planned Radiotherapy
  Arms: Consolidation radiotherapy
Radiation: Salvage Radiation — IMRT/VMAT technique. Patients receive radiotherapy once daily, 5 days a week for an average of 5 weeks. Radiotherapy is delivered to achieve a dosage of 49.22Gy/23f or 50Gy/25f to PGTV for lymphnode metastasis only patients and 40.66~49.22Gy/19f ~23f or 40~50Gy/20~25f for organ metastasis patients. Radiation treatment is planned after disease progression when recommended by multidisciplinary team.
  Other Names: Radiotherapy when needed
  Arms: Salvage radiotherapy

SUMMARY:
The treatment efficacy for stage IVb esophageal cancer has been improved through chemotherapy combined with immunotherapy recently.

On this basis, the investigators intend to conduct a prospective, multicenter phase II clinical trial to assess whether radiotherapy could further improve the survival of patients with metastatic esophageal cancer responding to PD-1 Inhibitor plus chemotherapy.

Accompanied tissue samples, blood samples and urine samples will be analyzed by molecular biological detection (Including Whole Exome Sequencing and proteomics) to explore potential biomarkers for predicting outcomes, efficacy and toxicity.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is one of the most common carcinomas with high morbidity and mortality worldwide. More than 30% of the patients were stage IV when diagnosed. Fluoropyrimidine plus platinum-based chemotherapy is recommended as first-line treatment for patients with metastatic EC for approximately four decades, however, only minimal improvement has been reached in overall survival (OS).

Recently, immune checkpoint inhibitors have shown effective antitumor activity in patients with unresectable, advanced or metastatic EC. Several randomized trials have demonstrated the PD-1 inhibitor could further improve the OS in patients with advanced esophageal squamous cell carcinoma (ESCC) on the basis of chemotherapy. Chemotherapy combined with immunotherapy has become one of the the standard treatment modality for metastatic EC.

As reported, for the patients with metastatic lung cancer or EC, locoregional radiotherapy could improve survival, especially in those who responding to systemic therapy. However, high-level evidence is still needed to assess whether these patients can benefit from local radiotherapy.

The efficacy of immunotherapy combined with chemotherapy is obviously better than that of chemotherapy alone. On this basis, locoregional radiotherapy may help those patients with metastatic EC responding to systemic therapy improve local control, relieve the local symptoms, and even improve survival.

Therefore, the investigators intend to conduct a prospective, multicenter phase II trial to assess the efficiency and safety of radiotherapy with chemotherapy and immunotherapy for patients with metastatic EC. Accompanied tissue samples, blood samples and urine samples will be analyzed by molecular biological detection to explore potential biomarkers for predicting outcomes, efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years, any gender
* 2. Histologically or cytologically confirmed squamous cell carcinoma of esophageal cancer. The initial clinical stage is IVb (2018 AJCC Cancer Staging Manual, 8th Edition) or recurrent patients with recurrence after radical treatment (radical treatment includes surgery and radiotherapy, but the recurrence site cannot be located in the previous radiotherapy field).
* 3. ECOG performance status <= 1. Patients aged 65 years and over need to complete G8 screening or Comprehensive Geriatric Assessment, and the final evaluation is good;
* 4.There was no significant abnormality in laboratory routine indicators such as blood routine and liver and kidney function;
* 5.For patients after definitive or preoperative radiotherapy, no recurrence was in the prior radiation filed;
* 6.Expected survival is more than 12 weeks;
* 7.Informed consent provided;
* 8.With response to 2-4 cycles of the first-line chemotherapy combined with immunotherapy.

Exclusion Criteria:

* 1.Patients with other cancer history except hypopharyngeal carcinoma in situ, non-malignant skin cancer and cervical carcinoma in situ.
* 2.Received surgery (except ostomy), chemotherapy or other anti-tumor treatment before enrollment；
* 3. Active infection currently exists . The following conditions occurred within 6 months before randomization: myocardial infarction, cerebrovascular accident, or received gastrointestinal, neurological, cardiopulmonary surgery;
* 4. History of allergy to chemotherapy drugs or autoimmune disease;
* 5. Participate in other clinical trials at present or within 4 weeks before enrollment;
* 6.There are factors such as high risk of fistula that radiotherapy cannot be safely carried out as assessed by the radiation oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity.
Enrollment: 120 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2028-10-26 (Estimated)

PRIMARY OUTCOMES:
EFFICACY:1-year overall survival probability | 12 month
  Overall survival was defined as the time from first dose to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported for all participants of the Intent-To-Treat (ITT) population. The Kaplan-Meier method was used to calculated the 1-year survival probability.

SECONDARY OUTCOMES:
EFFICACY: Median progression-free survival (PFS) | 12 month
  Median progression-free survival (PFS), was defined as the time from first dose to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first.
SAFETY: Acute toxicity rate | One month within the end of one specific treatment
  Acute toxicity Rate, was defined as the frequency of toxicities related to the treatment, which arises within one month after administration, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC AE5.0).
SAFETY: Late toxicity rate | One month after the end of one specific treatment.
  Late toxicity rate, was defined as the frequency of toxicities related to the treatment, which arises after one month after administration, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC AE5.0).
QUALITY OF LIFE: Change From Baseline in the EORTC QLQ-C30 Subscale Scores in Participants | 24 month
  The score of the participants evaluated by The EORTC core quality of life questionnaire (QLQ-C30). All of the scales and single-item measures range in score from 0 to100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning.
QUALITY OF LIFE: Change From Baseline in the EORTC QLQ-OES18 Subscale Scores in Participants | 24 month
  The score of the participants evaluated by The EORTC Quality of Life Questionnaire - Oesophageal Cancer Module (EORTC QLQ-OES18). All of the scales and single-item measures range in score from 0 to100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning.

OTHER OUTCOMES:
Biomarkers for the predicting of efficacy | 24 month
  To explore the dynamic changes of circulating tumor DNA (the frequency of specific mutations by Next-generation sequencing Methodology) from baseline, before and after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yang Liu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Zhi-Hao Lu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Cancer hospital, CAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in esophageal cancer. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact liuwenyang@cicams.ac.cn

REFERENCES:
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] Guttmann DM, Mitra N, Bekelman J, Metz JM, Plastaras J, Feng W, Swisher-McClure S. Improved Overall Survival with Aggressive Primary Tumor Radiotherapy for Patients with Metastatic Esophageal Cancer. J Thorac Oncol. 2017 Jul;12(7):1131-1142. doi: 10.1016/j.jtho.2017.03.026. Epub 2017 Apr 28. PMID 28461255